CLINICAL TRIAL: NCT03103568
Title: An Open-label, Non-randomized, 2-arm, 2-period Fixed Sequence Phase 1 Study to Evaluate the Potential Inhibition of Nitisinone on Cytochrome P450 2C9, 2D6, and 2E1 and the Organic Anion Transporters OAT1 and OAT3 in Healthy Volunteers
Brief Title: A Study to Investigate the Potential Influence of Nitisinone on the Metabolism and the Transport of Other Drugs in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Sobi.NTBC-006; 2016-004297-17 (EudraCT Number)
Record Dates: First submitted 2017-03-27; First posted 2017-04-06 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — nitisinone; Tolbutamide; Metoprolol; Chlorzoxazone; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - CYP substrates (Experimental): In Arm A of the clinical study the potential effect of multiple doses of nitisinone on the blood concentration of the active substances tolbutamide, metoprolol and chlorzoxazone will be investigated. These substances are metabolized by CYP2C9, CYP2D6 and CYP2E, respectively.
  A cocktail of the substances tolbutamide, metoprolol and chlorzoxazone will be given as a single dose at the beginning of the study and PK will be investigated. The participants will then administer nitisinone for two weeks until therapeutic serum concentrations level is reached. Serum and urine concentrations of nitisinone will then be investigated for 24 hours, followed by giving the substances tolbutamide, metoprolol and chlorzoxazone as a single dose together with nitisinone to investigate the PK during interaction.
  Interventions: Drug: Nitisinone in Arm A; Drug: Tolbutamide; Drug: Metoprolol; Drug: Chlorzoxazone
- Arm B - OAT substrates (Experimental): In Arm B of the clinical study the potential effect of multiple doses of nitisinone on the blood concentration of the active substances furosemide in the blood, which is transported by the transporter proteins OAT 1 and OAT 3, will be investigated.
  Furosemide will be given intravenously as a single dose at the beginning of the study and PK will be investigated. The participants will then administer nitisinone for two weeks until therapeutic dose is reached. Furosemide will then be given as a single dose together with nitisinone to investigate the PK during interaction.
  Interventions: Drug: Furosemide; Drug: Nitisinone in Arm B

INTERVENTIONS:
Drug: Nitisinone in Arm A — 4 capsules of 20 mg nitisinone (80 mg) is given once daily for 17 days.
  Other Names: Orfadin
  Arms: Arm A - CYP substrates
Drug: Tolbutamide — A 500 mg tablet is given as single oral dose 2 weeks apart.
  Arms: Arm A - CYP substrates
Drug: Metoprolol — A 50 mg tablet of metoprolol tartrate is given as single oral dose 2 weeks apart.
  Arms: Arm A - CYP substrates
Drug: Chlorzoxazone — A 250 mg tablet is given as single oral dose 2 weeks apart.
  Arms: Arm A - CYP substrates
Drug: Furosemide — A single intravenous dose of 20 mg administered as an i.v. infusion is given 2 weeks apart.
  Arms: Arm B - OAT substrates
Drug: Nitisinone in Arm B — 4 capsules of 20 mg nitisinone (80 mg) is given once daily for 16 days.
  Other Names: Orfadin
  Arms: Arm B - OAT substrates

SUMMARY:
An open-label, non-randomized, 2-arm, 2-period fixed sequence phase 1 study to evaluate the potential inhibition of nitisinone on cytochrome P450 2C9, 2D6, and 2E1 and the organic anion transporters OAT1 and OAT3 in healthy volunteers

DETAILED DESCRIPTION:
This is an open-label, non-randomized, 2-arm, 2-period fixed-sequence drug-drug interaction study in a total of 36 (18 in each arm) male and female healthy volunteers.

The study consists of: Screening, Period 1 (substrates only), Period 2 (substrates + nitisinone) and Follow-up. In the screening period, subjects will be assessed for eligibility. Eligible subjects will be assigned to one of two treatment arms. In Arm A, the potential inhibition of nitisinone on CYP2C9, CYP2D6, and CYP2E1 will be investigated. In Arm B, the possible combined effect of nitisinone on the renal transporters OAT1 and OAT3 will be investigated.

In Period 1, the subjects will receive a single dose of a CYP cocktail of 3 substrates (Arm A) or an OAT1/OAT3 substrate (Arm B). Substrate plasma concentrations will be measured for determination of substrate PK; for up to 48 hours in Arm A and for 8 hours in Arm B.

During Period 2, the treatment and assessments will vary slightly between the 2 treatment arms. Nitisinone will be administered for 14 days, without co-administration of any substrate, in order to reach steady state and the recommended target plasma concentration, before the interaction with the substrates is studied.

In Arm A, Period 2, subjects will receive nitisinone for 16 consecutive days (14 days on nitisinone only and two days on nitisinone + substrate). Nitisinone steady state PK will be determined based on plasma and urine samples collected during one dosage interval at steady state, on the day before co-administration of the substrates. Nitisinone will then be administered together with the CYP substrates, and plasma samples for determination of their PK will be collected as in Period 1. There will be a final nitisinone dose on the day after substrate administration in order to maintain therapeutic levels throughout the 48-hour sampling period.

In Arm B, Period 2, subjects will receive nitisinone for 15 consecutive days (14 days on nitisinone only and one day on nitisinone + substrate). No nitisinone steady state PK characterization will be conducted in this arm. On the last treatment day, the subjects will receive nitisinone together with the OAT1/OAT3 substrate. This will be followed by 8 hours of blood sampling for determination of substrate PK.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, 18 - 55 years of age inclusive, who are judged by the investigator to be healthy on the basis of a pre-study physical examination, which includes clinical chemistry, hematology and urinalysis, vital signs (pulse and blood pressure), and ECG.
2. Female subject must be either:

   a. Of none childbearing potential: i. post-menopausal (defined as at least 1 year without any menstruation without an alternative medical cause) , prior to Screening, or ii. documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening).

   b. Or, if of childbearing potential, i. must have a negative urine/serum pregnancy test at Screening, and ii. must be using highly effective methods of birth control [Acceptable forms of birth control include: 1) Placement of an intrauterine device (IUD) or intrauterine system (IUS). The devices must not release any hormones. (Note: The IUD must have a failure rate < 1 %) 2) the subject's male partner has undergone effective surgical sterilization before the female subject entered the clinical trial and he is the sole sexual partner of the female subject during the clinical trial. 3) Observe abstinence (acceptable only if it is the subject's usual lifestyle). ] (failure rate < 1% per year when used consistently and correctly) at least 3 months prior to Screening until 4 weeks after study termination in combination with an approved barrier method [Approved barrier methods of contraception include: condom (without spermicidal foam/gel/film/cream/suppository or fat- or oil-containing lubricants), or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.]. Women should be informed of the potential risks associated with becoming pregnant while enrolled.
3. Male subjects must agree to use a condom when having sexual intercourse with female partners of childbearing potential during treatment and up to 4 weeks after the last dose of study treatment.
4. Body weight 64 to 100 kg.
5. Body mass index (BMI) 18 - 30 kg/m2
6. Signed informed consent.

Exclusion Criteria:

1. Any medical condition which in the opinion of the investigator makes the subject unsuitable for inclusion.
2. Recent history or presence of clinically significant gastrointestinal, hepatic, renal, cardiovascular, hematological, metabolic, urological, pulmonary, neurological or psychiatric disorder.
3. History of hypoglycemia.
4. Current keratopathy, or other clinically relevant abnormalities, found by ophthalmologic slit-lamp examination.
5. Poor or ultra-rapid metabolism of CYP2D6 substrates confirmed by genotyping (exclusion criteria for Arm A only).
6. History of allergy, hypersensitivity or known contraindication to any of the drugs, or their excipients, used in this study.
7. History of sulfonamide allergy.
8. Continuous use of any non-topical medication within 1 month, over-the-counter preparations, herbal remedies , and all other medication within 14 days or less than 5 times the half-life of that medication, whichever is the longer, prior to first intake of an IMP.
9. Daily smoking > 10 cigarettes.
10. Daily consumption of more than 5 cups of coffee.
11. History of drug and/or alcohol abuse.
12. Positive drug screen or alcohol test.
13. Positive screens for HBsAg, anti-HCV, anti-HBc Ab, HepC, HIV 1 2 antibodies.
14. Pregnancy or breast feeding.
15. Female subjects using hormonal contraceptives.
16. Enrollment in another concurrent clinical study, or intake of an experimental drug, within 3 months prior to inclusion in this study.
17. Donation of more than 400 mL of blood within 90 days prior to drug administration or donation of more than 1.5 liters of blood in the 10 months prior to first intake of an IMP.
18. Foreseeable inability to cooperate with given instructions or study procedures.
19. Inability to give written informed consent or to comply fully with the protocol.
20. Vulnerable subjects, e.g., subjects kept in detention.
21. Soldiers, investigator, employees of the Sponsor or CRO.
22. Subject is not able to read, write and speak German.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) infinity for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  The primary outcome measure is to investigate the AUC for tolbutamide taken as a single dose with and without the presence of nitisinone.
AUC infinity for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  The primary outcome measure is to investigate the AUC for metoprolol taken as a single dose with and without presence of nitisinone.
AUC infinity for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  The primary outcome measure is to investigate the AUC for chlorzoxazone taken with and without the presence of nitisinone.
AUC infinity for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  The primary outcome measure is to investigate the AUC for furosemide with and without the presence of nitisinone.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  A secondary outcome measure is to investigate Cmax for tolbutamide taken as a single dose with and without the presence of nitisinone.
Time to maximum concentration (tmax) for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  A secondary outcome measure is to investigate tmax for tolbutamide taken as a single dose with and without the presence of nitisinone.
AUC last for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  A secondary outcome measure is to investigate AUC last for tolbutamide taken as a single dose with and without the presence of nitisinone.
Residual area for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  A secondary outcome measure is to investigate the residual area for tolbutamide taken as a single dose with and without the presence of nitisinone.
terminal half-life for CYP2C9 (tolbutamide) substrate | Blood samples will be obtained the following times in relation to tolbutamide administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose.
  A secondary outcome measure is to investigate the terminal half-life for tolbutamide taken as a single dose with and without the presence of nitisinone.
Cmax for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  A secondary outcome measure is to investigate Cmax for metoprolol taken as a single dose with and without the presence of nitisinone.
tmax for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  A secondary outcome measure is to investigate tmax for metoprolol taken as a single dose with and without the presence of nitisinone.
AUC last for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  A secondary outcome measure is to investigate AUClast for metoprolol taken as a single dose with and without the presence of nitisinone.
Residual area for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  A secondary outcome measure is to investigate the residual area for metoprolol taken as a single dose with and without the presence of nitisinone.
terminal half-life for CYP2D6 (metoprolol) substrate | Blood samples will be obtained the following times in relation to metoprolol administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9, 11, 15 and 23 h post-dose.
  A secondary outcome measure is to investigate the terminal half-life for metoprolol taken as a single dose with and without the presence of nitisinone.
Cmax for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  A secondary outcome measure is to investigate Cmax for chlorzoxazone taken as a single dose with and without the presence of nitisinone.
tmax for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  A secondary outcome measure is to investigate tmax for chlorzoxazone taken as a single dose with and without the presence of nitisinone.
AUC last for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  A secondary outcome measure is to investigate AUC last for chlorzoxazone taken as a single dose with and without the presence of nitisinone.
Residual area for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  A secondary outcome measure is to investigate the residual area for chlorzoxazone taken as a single dose with and without the presence of nitisinone.
terminal half-life for CYP2E1 (chlorzoxazone) substrate | Blood samples will be obtained the following times in relation to chlorzoxazone administration: predose and, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 7, 9 and 11 h post-dose.
  A secondary outcome measure is to investigate the terminal half-life for chlorzoxazone taken as a single dose with and without the presence of nitisinone.
Cmax for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  A secondary outcome measure is to investigate Cmax for furosemide taken as a single dose with and without the presence of nitisinone.
tmax for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  A secondary outcome measure is to investigate tmax for furosemide taken as a single dose with and without the presence of nitisinone.
AUC last for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  A secondary outcome measure is to investigate AUC last for furosemide taken as a single dose with and without the presence of nitisinone.
Residual area for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  A secondary outcome measure is to investigate the residual area for furosemide taken as a single dose with and without the presence of nitisinone.
terminal half-life for OAT1/OAT3 (furosemide) substrate | Blood samples will be obtained the following times in relation to furosemide administration: predose and, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 3, 4, 6, and 8 hours post-dose
  A secondary outcome measure is to investigate the terminal half-life for furosemide taken as a single dose with and without the presence of nitisinone.
24-hour plasma concentration profile for nitisinone at steady state. | Blood samples will be collected during 24 hours when steady state has been reached during the following time points: pre-dose and, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16 and 24 h postdose.
  A secondary outcome measure is to investigate the plasma concentration profile for nitisinone at steady state.
24 hour renal excretion for nitisinone at steady state. | Urine will be collected for 24 hours post nitisinone dosing and during the following time intervals: 0-3 hours, 3-6 hours, 6-9 hours, 9-12 hours and 12-24 hours.
  A secondary outcome measure is to investigate the urine excretion of nitisinone at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bröijersén, MD, PhD, Study Director — Swedish Orphan Biovitrum
Locations (1):
- PAREXEL EPCU Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No